CLINICAL TRIAL: NCT03189264
Title: Percutaneous Nephrolithotomy With Coaxial Dilatation vs Pneumatic Balloon for Treatment of Kidney Stones Greater Than 2 cm
Brief Title: Percutaneous Nephrolithotomy for Treatment of Kidney Stones Greater Than 2 cm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr Carlos Hernández (Other)
Responsible Party: Sponsor-Investigator, Dr Carlos Hernández, Urologist, Los Comuneros Hospital Universitario Bucaramanga
Organization: Los Comuneros Hospital Universitario Bucaramanga (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-05-08; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Renal Stone
Keywords: Percutaneous Nephrolithotomy; Postoperative Complications; Renal Stone; Surgical Success; Surgical Complications; Pneumatic Dilation
MeSH Terms: conditions — Nephrolithiasis; Postoperative Complications | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Percutaneous nephrolithotomy with Coaxial Dilatation (Active Comparator): Percutaneous nephrolithotomy with Coaxial Dilatation for treatment of kidney stones greater than 2 cm.
  Interventions: Procedure: percutaneous nephrolithotomy for kidney stones
- Percutaneous nephrolithotomy with Pneumatic Balloon (Placebo Comparator): Percutaneous nephrolithotomy with Pneumatic Balloon for treatment of kidney stones greater than 2 cm.
  Interventions: Procedure: percutaneous nephrolithotomy for kidney stones

INTERVENTIONS:
Procedure: percutaneous nephrolithotomy for kidney stones — Use of various methods of access to the renal collecting system (pneumatic balloon dilatation vs. traditional technique with coaxial dilators) during percutaneous nephrolithotomy for treatment of kidney stones greater than 2 cm.
  Other Names: Percutaneous nephrolithotomy with Coaxial Dilatation; Percutaneous nephrolithotomy with Pneumatic Balloon

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is a minimally invasive procedure considered as the treatment of choice for the management of large-scale and fully-formed kidney stones.This procedure has a 5% risk of complications including bleeding, the lesion of the collecting system, the risk of urinary infection and bacteremia. New surgical tools such as dilatation of the nephrostomy tract with mechanical dilatation contribute to the reduction of these risks, together with an improvement in the operative times and a lower rate of complications.

At present there are multiple scales measuring the lithiasic morphology (Guy, the STONE nephrolitometry score system and the nomogram of the Office of Clinical Investigation of the Endourology Society - CROES) which allow to evaluate the degree of complexity of the stone, the possibility of residual stones and the risk of complications. These tools allow us to do a better analysis of the risk factors of the patient who will be taken to this type of endoscopic procedure in order to decrease morbidity and complication rates.

Hypothesis:

The use of pneumatic dilators during percutaneous nephrolithotomy reduces the rates of intraoperative and postoperative complications, which would have an impact on hospitalization times and surgical success for the management of renal stone.

DETAILED DESCRIPTION:
Nephrolithiasis is a major worldwide source of morbidity, constituting a common urological disease affecting 10-15% of the world population, with a subsequent clinical relapse rate of approximately 50%. Recent technological and surgical advances have reduced the need for open surgery with less invasive procedures, such as percutaneous nephrolithotomy (PCNL), extracorporeal shock wave lithotripsy (SWL) and retrograde ureteroscopy. The selection of the surgical procedure generally depends on the size, composition, location of the renal stone, the existence of obstruction and anatomical variations of the urinary system. Today, PCNL is the established procedure for stone greater than 2 cm; The procedure usually involves three main stages: it begins with the insertion of a ureteral catheter to perform a retrograde study with contrast medium where the anatomy of the kidney is evaluated, then the puncture is performed by inserting a surgical needle on the skin to the specific location of the stone, with subsequent dilatation of the tract to the collecting system, and once this access has been made it is proceeded to carry out the fragmentation and extraction of the stone through various types of instruments.

The success and results of the treatment of surgery are very well known and highly dependent on precision in the puncture stage (the stones must be achieved with a precise and direct path), make this step is the most challenge for surgeons. The ideal access is one that allows complete removal of the stones while minimizing intraoperative bleeding. Needle punctures and their complications, such as kidney injuries and adjacent organs, eventually impair the overall surgical success and outcome of the patient. Although PCNL is considered minimally invasive surgery (MIS) with many associated benefits, such as the production of small incisions in the patient, reducing hospitalization time and postoperative recovery, some complications still occur frequently. The dilation of the nephrostomy tract is the second step in which there are more complications, since it depends on an optimal puncture of the collecting system and a precise manual control to avoid damages of the collecting system or to increase the risks of bleeding.

Restricted vision, difficulty in handling the Instrumental, restrictive mobility within the kidney, skill levels of hand-eye coordination of the surgeon, deviation of the needle, moving anatomical objective, are a constant challenge for the surgeon. Several technological advances have been proposed to improve the effectiveness of this procedure. In regard to puncture and dilatation, relevant contributions have been provided by the improvement in medical imaging techniques, as well as the fusion of multiple imaging procedures.

Main goal

To determine the highest rate of intraoperative and early postoperative complications (bleeding, pain) with the use of the various methods of access to the renal collecting system during percutaneous nephrolithotomy for the treatment of kidney stones greater than 2 cm than 2 cm between April 2017 and January 2018.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Non-staghorn kidney stones greater than 2 cm

Exclusion Criteria:

* Coagulopathies
* Solitary Functioning Kidney
* Pyonephrosis
* Pregnancy
* Urinary tract infection
* Cardiopulmonary Restrictions Limiting Prone Position
* BMI greater than 35
* More of 2 puncture of the excretory tract
* STONE score equal or greater than 12

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of intraoperative and postoperative complications that occur with the use of pneumatic dilation and with traditional coaxial dilatation. | 8 weeks
  To determine the highest rate of intraoperative and early postoperative complications with the use of various methods of access to the renal collecting system during percutaneous nephrolithotomy for the treatment of kidney stones greater than 2 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Hernandez, MD, Principal Investigator — HOSPITAL UNIVERSITARIO LOS COMUNEROS; Andres Gutierrez, MD, Study Chair — HOSPITAL UNIVERSITARIO LOS COMUNEROS; Jose G Ramos, MD, Study Chair — HOSPITAL UNIVERSITARIO LOS COMUNEROS; Diana M Chaparro, MD, Study Chair — HOSPITAL UNIVERSITARIO LOS COMUNEROS; Eduardo Ardila, MD, Study Chair — HOSPITAL UNIVERSITARIO LOS COMUNEROS
Locations (1):
- Hospital Universitario Los Comuneros, Bucaramanga, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopes T, Sangam K, Alken P, Barroilhet BS, Saussine C, Shi L, de la Rosette J; Clinical Research Office of The Endourological Society Percutaneous Nephrolithotomy Study Group. The Clinical Research Office of the Endourological Society Percutaneous Nephrolithotomy Global Study: tract dilation comparisons in 5537 patients. J Endourol. 2011 May;25(5):755-62. doi: 10.1089/end.2010.0488. Epub 2011 Mar 9. PMID 21388242
- [Result] GOODWIN WE, CASEY WC, WOOLF W. Percutaneous trocar (needle) nephrostomy in hydronephrosis. J Am Med Assoc. 1955 Mar 12;157(11):891-4. doi: 10.1001/jama.1955.02950280015005. No abstract available. PMID 13233046
- [Result] Fernstrom I, Johansson B. Percutaneous pyelolithotomy. A new extraction technique. Scand J Urol Nephrol. 1976;10(3):257-9. doi: 10.1080/21681805.1976.11882084. PMID 1006190
- [Result] Beiko D, Elkoushy MA, Kokorovic A, Roberts G, Robb S, Andonian S. Ambulatory percutaneous nephrolithotomy: what is the rate of readmission? J Endourol. 2015 Apr;29(4):410-4. doi: 10.1089/end.2014.0584. Epub 2014 Oct 23. PMID 25221917
- [Result] Tailly T, Razvi H. The S.T.O.N.E. nephrolithometry scoring system: How valid is it? Can Urol Assoc J. 2015 May-Jun;9(5-6):196. doi: 10.5489/cuaj.3020. No abstract available. PMID 26225169
- [Result] Thomas K, Smith NC, Hegarty N, Glass JM. The Guy's stone score--grading the complexity of percutaneous nephrolithotomy procedures. Urology. 2011 Aug;78(2):277-81. doi: 10.1016/j.urology.2010.12.026. Epub 2011 Feb 17. PMID 21333334
- [Result] Akhavein A, Henriksen C, Syed J, Bird VG. Prediction of single procedure success rate using S.T.O.N.E. nephrolithometry surgical classification system with strict criteria for surgical outcome. Urology. 2015 Jan;85(1):69-73. doi: 10.1016/j.urology.2014.09.010. PMID 25530366
- [Result] Okhunov Z, Friedlander JI, George AK, Duty BD, Moreira DM, Srinivasan AK, Hillelsohn J, Smith AD, Okeke Z. S.T.O.N.E. nephrolithometry: novel surgical classification system for kidney calculi. Urology. 2013 Jun;81(6):1154-9. doi: 10.1016/j.urology.2012.10.083. Epub 2013 Mar 26. PMID 23540858
- [Result] Shahrour W, Andonian S. Ambulatory percutaneous nephrolithotomy: initial series. Urology. 2010 Dec;76(6):1288-92. doi: 10.1016/j.urology.2010.08.001. PMID 21130245
- [Result] Beiko D, Lee L. Outpatient tubeless percutaneous nephrolithotomy: the initial case series. Can Urol Assoc J. 2010 Aug;4(4):E86-90. doi: 10.5489/cuaj.886. PMID 20694090